CLINICAL TRIAL: NCT03187951
Title: PancFit: Multimodal Exercise During Preoperative Therapy for Pancreatic Cancer: A Randomized Trial Testing Effects on Fitness, Health-Related Quality of Life, and Tumor Vasculature
Brief Title: PancFit: Multimodal Exercise During Preoperative Therapy for Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0198; NCI-2018-01183 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Other Disorders of Glucose Regulation and Pancreatic Internal Secretion; Pancreatic Cancer
Keywords: Other disorders of glucose regulation and pancreatic internal secretion; Pancreatic cancer; Questionnaires; Surveys; Nutritional Questionnaire; Nutritional Counseling; Booklet; Pamphlet; Educational materials; Aerobic Exercise; Strength Training Exercises; Physical Assessments; Walk Test
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires; Nutrition Assessment; Exercise; Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Standard of Care (SOC) (Experimental): After completion of chemotherapy and/or radiation, 3-6 weeks after surgery, and then 3-7 months after surgery: Participants complete 4 questionnaires about physical abilities, motivation, and quality of life. Participant's hand grip strength measured. Participants arm strength measured using an arm curl test. Participants asked to rise from a chair without using their arms to push off. Participants complete a 6-minute walk test to see how far participant can walk in 6 minutes. Participants complete a nutritional questionnaire and receive nutritional counseling. Participants receive educational materials and personalized counseling based on participant's answers.
  Participants encouraged to remain active during chemotherapy and/or radiation. Participants receive a booklet that contains a stretching guide with full-body stretches and safety.
  Interventions: Behavioral: Questionnaires; Behavioral: Nutritional Questionnaire and Nutritional Counseling; Other: Booklet; Behavioral: Physical Assessments
- Arm B: Multi-Modal Exercise and Nutrition Program (MMENP) (Experimental): After completion of chemotherapy and/or radiation, 3-6 weeks after surgery, then 3-7 months after surgery: Participants complete 4 questionnaires about physical abilities, motivation, and quality of life. Participant's hand grip strength measured. Participants arm strength measured. Participants asked to rise from a chair without using their arms to push off. Participants complete a 6-minute walk test to see how far participant can walk in 6 minutes. Participants complete a nutritional questionnaire and receive nutritional counseling. Participants receive educational materials and personalized counseling based on participant's answers.
  Participants complete moderate-intensity aerobic exercise 5 days each week. Participants complete strength training exercises 2 times per week.
  Participants contacted by phone by member of study staff 1 time each week for the first 4 weeks, and then every 2 weeks after that for behavioral skills training and to see how participant is doing.
  Interventions: Behavioral: Questionnaires; Behavioral: Nutritional Questionnaire and Nutritional Counseling; Behavioral: Aerobic Exercise and Strength Training Exercises; Behavioral: Phone Calls; Behavioral: Physical Assessments

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete 4 questionnaires about physical abilities, motivation, and quality of life They should take about 25 minutes total to complete.
  Other Names: Surveys
Behavioral: Nutritional Questionnaire and Nutritional Counseling — Participants complete a nutritional questionnaire and receive nutritional counseling. It should take about 5 minutes to complete. Participants receive educational materials and personalized counseling based on participant's answers.
Other: Booklet — Participants receive a booklet that contains a stretching guide with full-body stretches and safety.
  Other Names: Pamphlet; Educational materials
  Arms: Arm A: Standard of Care (SOC)
Behavioral: Aerobic Exercise and Strength Training Exercises — Participants complete up to 30 minutes of moderate-intensity aerobic exercise (such as brisk walking, stationary cycling, and/or elliptical or stair stepping machines) for at least 5 days each week. Participants complete strength training exercises at least 2 times per week.
  Arms: Arm B: Multi-Modal Exercise and Nutrition Program (MMENP)
Behavioral: Phone Calls — Participants contacted by phone by member of study staff one (1) time each week for the first 4 weeks, and then every 2 weeks after that for behavioral skills training and to see how participant is doing. These calls should last about 15 minutes.
  Arms: Arm B: Multi-Modal Exercise and Nutrition Program (MMENP)
Behavioral: Physical Assessments — After completion of chemotherapy and/or radiation, 3-6 weeks after surgery, and then 3-7 months after surgery: Participant's hand grip strength measured using a hand-held machine. Participants arm strength measured using an arm curl test. Participants asked to rise from a chair without using their arms to push off. Participants complete a 6-minute walk test to see how far participant can walk in 6 minutes.

SUMMARY:
Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this clinical research study is to learn if regular exercise and behavioral skills training can help to improve physical activity in patients with pancreatic cancer who are scheduled to receive chemotherapy and/or radiation before standard-of-care surgery.

This is an investigational study.

Up to 128 participants will be enrolled on this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study arms. This is done because no one knows if one study arm is better than, the same, or worse than the other group.

If you are in Arm A, you will not take part in a structured exercise program. If you are in Arm B, you will take part in a structured exercise program and behavioral skills training as described below.

Length of Study:

You will continue to take part in this study for up to 7 months after your scheduled standard-of-care surgery. However, if intolerable side effects occur or the disease appears to get worse, the study staff will decide if continuing the exercise program is in your best interest.

Study Visits:

At your baseline visit, after you complete chemotherapy and/or radiation, 3-6 weeks after surgery, and then 3-7 months after surgery:

* You will complete 4 questionnaires about your physical abilities, motivation, and quality of life. They should take about 25 minutes total to complete.
* Your hand grip strength will be measured using a hand-held machine
* Your arm strength will be measured using an arm curl test. You will be given a small weight (about 5-8 pounds) and asked to perform as many bicep curls as you can for 30 seconds.
* You will be asked to rise from a chair without using your arms to push off.
* You will complete a 6-minute walk test to see how far you can walk in 6 minutes.
* You will complete a nutritional questionnaire and receive nutritional counseling. The questionnaire will ask about your diet and any recent weight loss. It should take about 5 minutes to complete. After you complete the questionnaire, you will receive educational materials and personalized counseling based on your answers.
* If you are in Arm B, you will receive behavioral skills training to teach you ways to monitor your health, set goals, and reward yourself. It should take about 15 minutes to complete.
* At the baseline visit, you will be given a Fitbit Charge 2 activity tracker to wear during the study. This is a small device designed to record your physical activity and sleep during the study. This device will allow you to monitor your own physical activity and sleep and may help you achieve your goals. You can keep the Fitbit after the study is over.

If you are in Arm B, one (1) time each week for the first 4 weeks and then every 2 weeks after that, a member of the study staff will contact you by phone for behavioral skills training and to see how you are doing. These calls should last about 15 minutes.

For 2 weeks during each phase of chemotherapy and/or radiation you receive, you will wear a small activity monitor on an elastic band. This will be worn in addition to your Fitbit.

Exercise Programs:

ARM A:

If you are in Arm A, you will be encouraged to remain active during chemotherapy and/or radiation, but you will not receive instruction about aerobic or strengthening exercises. You will receive a booklet that contains a stretching guide with full-body stretches and safety.

ARM B:

If you are in Arm B, you will be asked to complete up to 30 minutes of moderate-intensity aerobic exercise (such as brisk walking, stationary cycling, and/or elliptical or stair stepping machines) for at least 5 days each week.

You will also complete strength training exercises at least 2 times per week. You will complete 1 set of 10-15 repetitions for each of the 8 exercises that you are taught. Over time, the amount of resistance, repetitions, and/or sets may increase or decrease based on your strength. You will be given 5 different resistance tubes to complete these exercises, but you may use free-weights or machines if you prefer.

You should complete warm up exercises and 5 minutes of stretching before and after strength training.

You must keep a daily activity log to document your exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Pancreatic cancer of any type, biopsy-proven
2. Scheduled to receive preoperative therapy (chemotherapy, radiation or chemoradiation) either on- or off-protocol.
3. Anticipated to undergo pancreatectomy in >/= 6 weeks from enrollment
4. Able to understand the description of the study and willing to participate
5. Able to understand the exercise program
6. Able to maintain daily exercise logs
7. Telephone or email access and agreement to engage with the research personnel via phone or email
8. Meet all screening requirements.

Exclusion Criteria:

1. Non-English speaking
2. Unable to complete the baseline assessment questionnaires or functional assessments
3. Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV)
4. Recent fracture or acute musculoskeletal injury that precludes the ability to weight bear fully on all 4 limbs in order to participate in an exercise intervention
5. Numeric pain rating scale of >/= 7 out of 10
6. Myopathic or rheumatologic disease that impacts physical function
7. Recurrent cancer following prior resection
8. Neuroendocrine cancer
9. Completed preoperative therapy and are on their presurgical rest period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test (6MWT) | Change compared from baseline to date surgery is scheduled
  Primary endpoint is the change in 6MWT distance, measured in meters, between the time at which preoperative therapy is administered (T0) and the time at which it ends (T1).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Katz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ngo-Huang AT, Parker NH, Xiao L, Schadler KL, Petzel MQB, Prakash LR, Kim MP, Tzeng CD, Lee JE, Ikoma N, Wolff RA, Javle MM, Koay EJ, Pant SD, Folloder JP, Wang X, Cotto AM, Ju YR, Garg N, Wang H, Bruera ED, Basen-Engquist KM, Katz MHG. Effects of a Pragmatic Home-based Exercise Program Concurrent With Neoadjuvant Therapy on Physical Function of Patients With Pancreatic Cancer: The PancFit Randomized Clinical Trial. Ann Surg. 2023 Jul 1;278(1):22-30. doi: 10.1097/SLA.0000000000005878. Epub 2023 Apr 7. PMID 37026453
- See also: MD Anderson Cancer Center — http://www.mdanderson.org